CLINICAL TRIAL: NCT02550431
Title: Trans Health: Evaluation of Markers of Cardio-metabolic Health and Well-being in Transgender Youth
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1215; UL1TR001082 (NIH)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Transgendered Persons

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This study plans to learn more about puberty blockers and cross (testosterone and estradiol). There is not much known about how these medications affect hormone levels, heart health and overall general health in young transgender individuals.

DETAILED DESCRIPTION:
This study plans to learn more about puberty blockers and cross (testosterone and estradiol). There is not much known about how these medications affect hormone levels, heart health and overall general health in young transgender individuals.

ELIGIBILITY:
Inclusion Criteria:

* Followed in Endocrinology Clinic or Adolescent Medicine Clinic at Children's Hospital Colorado
* Between age 9 and 21 years (inclusive)
* Identifies as transgender
* Has been on pubertal blockade or cross-sex hormones for at least three months.

Exclusion Criteria:

* Known diabetes
* Presence of significant medical or psychiatric comorbidities
* Using hormones not prescribed by a physician

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Transgender youth ages 9 to 21 years of age who have been on a Gonadotropin-releasing hormone (GnRH) agonist or cross-sex hormones for at least three months
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Reproductive hormone concentrations in transgender youth on cross-sex hormones and/or puberty blockers and compared to age-, natal sex- and body mass index (BMI)-matched controls. | at enrollment
Markers of cardiometabolic risk in transgender youth on cross-sex hormones and/or puberty blockers and compared to age-, natal sex- and BMI-matched controls | at enrollment
Body composition as measured by Dual-energy X-ray absorptiometry (DEXA) in transgender youth compared to age- and BMI-matched controls of both sexes. | at enrollment
Data on quality of life as measured by the Pediatric Quality of Life Inventory (PedsQL) compared to published norms | at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Natalie J Nokoff, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Nokoff NJ, Scarbro SL, Moreau KL, Zeitler P, Nadeau KJ, Reirden D, Juarez-Colunga E, Kelsey MM. Body Composition and Markers of Cardiometabolic Health in Transgender Youth on Gonadotropin-Releasing Hormone Agonists. Transgend Health. 2021 Apr 16;6(2):111-119. doi: 10.1089/trgh.2020.0029. eCollection 2021 Apr. PMID 33937527
- [Derived] Nokoff NJ, Scarbro SL, Moreau KL, Zeitler P, Nadeau KJ, Juarez-Colunga E, Kelsey MM. Body Composition and Markers of Cardiometabolic Health in Transgender Youth Compared With Cisgender Youth. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e704-14. doi: 10.1210/clinem/dgz029. PMID 31544944